CLINICAL TRIAL: NCT00059787
Title: Phase II Study of Erlotinib Plus Carboplatin and Paclitaxel in Patients With Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Erlotinib Plus Carboplatin and Paclitaxel in Ovarian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00026; NYU 02-30 (Other: New York University); N01CM62204 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2013-05

CONDITIONS: Brenner Tumor; Fallopian Tube Cancer; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Taxes; Carboplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel, carboplatin, erlotinib (Experimental): Carboplatin and paclitaxel IV every 21 days x 6 cycles plus oral erlotinib
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: erlotinib

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: erlotinib — Given PO
  Other Names: CP-358,774; OSI-774

SUMMARY:
This phase II trial is studying the side effects of giving erlotinib together with carboplatin and paclitaxel and to see how well it works in treating patients with stage III or stage IV ovarian, fallopian tube, or primary peritoneal cancer. Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy such as carboplatin and paclitaxel use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish whether the addition of OSI-774 (Tarceva) to the combination of paclitaxel and carboplatin encourages pathologic complete response (pCR) rates in patients with Stage III optimally cytoreduced (stratum 1) and Stage III suboptimally cytoreduced or Stage IV (stratum 2) ovarian, primary peritoneal or fallopian tube carcinomas when used as front line therapy.

II. To determine the degree and type of toxicity associated with this combined regimen.

SECONDARY OBJECTIVES:

I. To establish baseline epidermal growth factor receptor (EGFR), truncated EGFR (EGFRvIII), phosphorylated EGFR (pEGFR) and related signal transduction pathway protein expression levels (such as the mitogen activated protein kinase p-ERK, AKT phosphorylation and Her2/neu) in tumor samples obtained pretreatment, and to correlate these with achieving pCR.

II. To describe changes in EGFR, EGFRvIII, pEGFR expression levels and other related signal transduction pathway expression occurring during treatment with OSI-774 in combination with chemotherapy.

III. To determine the effect of the addition of OSI-774 (Tarceva) to the combination of paclitaxel and carboplatin on progression-free interval in patients with Stage III optimally cytoreduced (stratum 1) and Stage III suboptimally cytoreduced or Stage IV (stratum 2) ovarian or primary peritoneal carcinomas when used as front line therapy.

IV. To determine the tolerability of twelve months of maintenance treatment with OSI-774 for patients achieving pCR, and to measure the progression-free interval for this population.

V. To document cutaneous effects of OSI 774 prospectively, and to correlate the degree of skin rash with clinical and translational endpoints.

OUTLINE: This is a non-randomized study. Patients are stratified according to disease stage (stage III with optimal residual disease vs stage III with suboptimal residual disease or stage IV).

Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive oral erlotinib daily. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a pathologic complete response, those initially suboptimally debulked with a response, and patients who elect not to undergo surgical reassessment but who achieve a complete clinical response receive maintenance erlotinib for an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of primary peritoneal carcinoma, fallopian tube epithelial ovarian carcinoma, Stage III with either greater than 1 cm (suboptimal) residual disease following initial surgery, or Stage IV; all patients must either have had appropriate surgery for ovarian, fallopian tube or peritoneal carcinoma with appropriate tissue available for histologic evaluation to confirm diagnosis and stage or must be unresectable at time of diagnosis (to be determined by gynecological oncologist); cytology alone is not adequate
* Patients with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (NOS)
* Patients must begin chemotherapy on this study no more than twelve weeks postoperatively
* Patients must not have received chemotherapy within five years prior to enrollment
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Neuropathy (sensory and motor) =< CTC grade 1
* No medical contraindications to planned regimen
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had courses of chemotherapy within the five years prior to entering the study
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition OSI-774 or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because OSI-774 has the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with OSI-774, breastfeeding should be discontinued if the mother is treated with OSI-774; these potential risks may also apply to other agents used in this study
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with OSI-774 or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Blank, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Blank SV, Christos P, Curtin JP, Goldman N, Runowicz CD, Sparano JA, Liebes L, Chen HX, Muggia FM. Erlotinib added to carboplatin and paclitaxel as first-line treatment of ovarian cancer: a phase II study based on surgical reassessment. Gynecol Oncol. 2010 Dec;119(3):451-6. doi: 10.1016/j.ygyno.2010.08.008. Epub 2010 Sep 15. PMID 20837357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 patients were enrolled between June 2003 and December 2006.
Groups:
- Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Patients also receive oral erlotinib daily. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a pathologic complete response, those initially suboptimally debulked with a response, and patients who elect not to undergo surgical reassessment but who achieve a complete clinical response receive maintenance erlotinib for an additional 12 months.
  paclitaxel: Given IV
  carboplatin: Given IV
  erlotinib hydrochloride: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Started | 56
Completed | 36
Not Completed | 20
Not completed — Adverse Event | 13
Not completed — disease progression | 2
Not completed — ineligible | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 55.5 [22 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 2
  Asian | 5
  White | 42
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rates
Description: Pathologic complete response was defined as having no pathologic or cytologic evidence of disease following surgical reassessment.
Time Frame: Up to 7 years
Population: Patients who had optimally debulking surgery
Measure: Number; unit: participants
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Number analyzed (Participants) | 28
participants | 8

2. Primary Outcome: The Percentage of Participants Experiencing Toxicty (Grade 2 and Grade 3/4) Associated With the Combined Regimen
Description: Adverse event assessment
Time Frame: For the duration of the study up to 7 years
Population: Patients enrolled on all stratums included
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel, Carboplatin, Erlotinib
Number analyzed (Participants) | 56
percentage of participants
  Grade 3-4 neutropenia | 18
  Grade 3-4 skin rash | 17
  Grade 3-4 thrombocytopenia | 7
  Grade 3-4 infection | 7
  Grade 3-4 fatigue | 5
  Grade 3 diarrhea | 4
  Grade 2 skin rash | 21
  Grade 2 diarrhea | 7

3. Secondary Outcome: To Measure EGFR Gene Amplification in Tumor Specimens
Time Frame: The duration of the study for up to 7 years
Population: Tumor specimens were evaluated for EGFR gene amplification in 20 patients
Measure: Number; unit: number of tumor specimens
Arm/Group | Paclitaxel, Carboplatin, Erlotinib
Number analyzed (Participants) | 20
number of tumor specimens
  No amplification | 11
  Low-level amplification | 6
  moderate high amplification | 3

4. Secondary Outcome: To Determine Progession Free Survival With the Addition of OSI-774 (Tarceva) to the Combination of Paclitaxel and Carboplatin
Time Frame: The duration of the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Number analyzed (Participants) | 51
months | 34.3 [23.9 to 51.8]

5. Secondary Outcome: To Determine the Tolerability of Twelve Months of Maintenance Treatment
Time Frame: Twelve months of maintenance
Measure: Number; unit: participants
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Number analyzed (Participants) | 16
participants
  No recurrence | 12
  Recurrence | 4

ADVERSE EVENTS:
Arm/Group | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 20/56
Other Adverse Events (participants affected / at risk) | 17/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride) (N=56)
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Infection (Infections and infestations) | 4
Rash: desquamation (Skin and subcutaneous tissue disorders) | 9
Fatigue (General disorders) | 3
Alanine transaminase (Hepatobiliary disorders) | 1
Aspartate transaminase (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Erlotinib Hydrochloride) (N=56)
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 13
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 12
Nausea (General disorders) | 10
Rash: desquamation (Skin and subcutaneous tissue disorders) | 17
Mucositis: oral (Gastrointestinal disorders) | 6
Neuropathy (Nervous system disorders) | 12
Pain: abdomen (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less